CLINICAL TRIAL: NCT00348712
Title: Efficacy and Safety of Inhaled Pre-prandial Human Insulin Plus Metformin Versus Rosiglitazone Plus Metformin in Type 2 Diabetes
Brief Title: Efficacy and Safety of Inhaled Pre-prandial Human Insulin in Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1390; 2006-000796-15 (EudraCT Number)
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: inhaled human insulin; Drug: metformin
- B (Active Comparator)
  Interventions: Drug: rosiglitazone; Drug: metformin

INTERVENTIONS:
Drug: rosiglitazone — Tablets, 4 mg once or twice daily.
  Arms: B
Drug: inhaled human insulin — Treat-to-target dose titration scheme, inhalation.
  Other Names: NN1998
  Arms: A
Drug: metformin — Tablets, 2000 mg/day.

SUMMARY:
This trial is conducted in Europe.

The aim of this research study is to compare the efficacy of adding inhaled preprandial insulin to metformin compared to adding rosiglitazone to metformin for the treatment of type 2 diabetes and to verify its safety (hypoglycaemia, pulmonary function, body weight, insulin antibodies and side effects).

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treated with OAD(s) for more than or equal to 2 months
* Body mass index of (BMI) less than or equal to 40.0 kg/m2
* HbA1c greater than or equal to 7.5% and less than or equal to 11.0 % for subjects in OAD monotherapy and HbA1c greater than or equal to 7.0% and less than or equal to 10.0 % for subjects on OAD combination therapy

Exclusion Criteria:

* Recurrent major hypoglycaemia
* Current smoking or smoking within the last 6 months
* Impaired hepatic or renal function
* Cardiac disorders
* Uncontrolled hypertension
* Proliferative retinopathy or maculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2006-10-30 (Actual); Primary Completion 2008-03-05 (Actual); Study Completion 2008-03-05 (Actual)

PRIMARY OUTCOMES:
Treatment difference in HbA1c | After 26 weeks

SECONDARY OUTCOMES:
Adverse events | For the duration of the trial
Body weight | For the duration of the trial
Lung function | For the duration of the trial
Blood glucose | For the duration of the trial
Hypoglycaemia | For the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (70):
- Austria (2):
  - Novo Nordisk Investigational Site, Ebreichsdorf
  - Novo Nordisk Investigational Site, Vienna
- Finland (3):
  - Novo Nordisk Investigational Site, Joensuu
  - Novo Nordisk Investigational Site, Kirkkonummi
  - Novo Nordisk Investigational Site, Turku
- France (11):
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Mougins
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Pessac
  - Novo Nordisk Investigational Site, Pointe à Pitre
  - Novo Nordisk Investigational Site, Roubaix
  - Novo Nordisk Investigational Site, Tours
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (19):
  - Novo Nordisk Investigational Site, Aschaffenburg
  - Novo Nordisk Investigational Site, Augsburg
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Darmstadt
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Flörsheim
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Fulda
  - Novo Nordisk Investigational Site, Genthin
  - Novo Nordisk Investigational Site, Hermaringen
  - Novo Nordisk Investigational Site, Kutenholz-Mulsum
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Pirna
  - Novo Nordisk Investigational Site, Schkeuditz
  - Novo Nordisk Investigational Site, Wangen
  - Novo Nordisk Investigational Site, Wiesbaden
- Ireland (2):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Waterford
- Netherlands (7):
  - Novo Nordisk Investigational Site, Delft
  - Novo Nordisk Investigational Site, Drachten
  - Novo Nordisk Investigational Site, Rijswijk
  - Novo Nordisk Investigational Site, Roelofarendsveen
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Vlodrop
  - Novo Nordisk Investigational Site, Zwijndrecht
- Spain (10):
  - Novo Nordisk Investigational Site, Alzira
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Gijón
  - Novo Nordisk Investigational Site, Majadahonda
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Partida de Bacarot
  - Novo Nordisk Investigational Site, Pontevedra
  - Novo Nordisk Investigational Site, Reus
  - Novo Nordisk Investigational Site, San Juan
  - Novo Nordisk Investigational Site, Seville
- Switzerland (3):
  - Novo Nordisk Investigational Site, Interlaken-Unterseen
  - Novo Nordisk Investigational Site, Olten
  - Novo Nordisk Investigational Site, Zurich
- United Kingdom (13):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bradford-on-Avon
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Trowbridge
  - Novo Nordisk Investigational Site, Wirral, Merseyside
  - Novo Nordisk Investigational Site, York

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com